CLINICAL TRIAL: NCT04857398
Title: A Trial Investigating the Pharmacokinetic Properties of Insulin Icodec in Chinese Subjects With Type 2 Diabetes
Brief Title: A Study to Test How a New Long-acting Insulin (Insulin Icodec) Works in the Body of People From China With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4571; U1111-1244-4473 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-04-22; First posted 2021-04-23 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin icodec (Experimental): The participants will receive an individualised weekly dose of subcutaneously (s.c.) insulin icodec for 6 weeks
  Interventions: Drug: insulin icodec

INTERVENTIONS:
Drug: insulin icodec — Participants will get insulin icodec once a week for 6 weeks. The medicine will be injected under the skin.
  The study will last for 15 to 22 weeks.

SUMMARY:
This study is looking at the way insulin icodec stays and moves over time in the blood after injections in Chinese people with type 2 diabetes.

Participants will get insulin icodec once a week for 6 weeks. The medicine will be injected under the skin of the thigh. There will also be a run-in period that will last between 1 week and 8 weeks with daily doses of insulin degludec before start on insulin icodec.

The study will last for about 15 to 22 weeks. Participants will have about 17 visits with the study doctor including phone contact during your run-in period.

Participants will have blood samples taken at the clinic visits. Several samples of participants blood will be taken for up to 48 hours after getting the first and the last dose of insulin icodec.

Participants must be a Chinese person diagnosed with type 2 diabetes for at least 6 months and be on basal insulin treatment for at least 2 months before participating in the study.

Women: Women cannot take part if pregnant, breast-feeding or plan to become pregnant during the study period

ELIGIBILITY:
Inclusion Criteria:

* Chinese male or female
* Aged 18-64 years (both inclusive) at the time of signing informed consent
* Body mass index between 18 and 38 kg/m^2 (both inclusive)
* HbA1c (glycated haemoglobin) below or equal to 9% at screening
* Current daily basal insulin treatment greater than or equal to 0.2 (I)U/kg/day greater than or equal to 60 days prior to the day of screening with or without any of the following anti-diabetic drugs/regimens with stable doses greater than or equal to 60 days prior to the day of screening:
* Any metformin formulation
* Other oral antidiabetic drugs: DPP-4 (Dipeptidyl-peptidase-4) Inhibitors , SGLT2 (Sodium-glucose co-transporter-2) inhibitors, Oral combination products (for the allowed individual oral antidiabetic drugs)
* Oral or injectable GLP-1 (Glucagon Like Peptide 1) Receptor Agonists

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measures as required by local regulation or practice).
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days prior to screening or in the period between screening and run-in. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event within the past 180 days) or hypoglycaemic unawareness as judged by the investigator or hospitalisation for diabetic ketoacidosis within the past 180 days prior to the day of screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin icodec concentration-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (Day 36)
  pmol*h/L

SECONDARY OUTCOMES:
Area under the serum insulin icodec concentration-time curve during one dosing interval at steady state divided by dose | From 0 to 168 hours after trial product administration (Day 36)
  (pmol*h/L)/(U/kg)
Maximum observed serum insulin icodec concentration after the last dose | From 0 to 168 hours after trial product administration (Day 36)
  pmol/L
Maximum observed serum insulin icodec concentration after the last dose divided by dose | From 0 to 168 hours after trial product administration (Day 36)
  (pmol/L)/(U/kg)
Time to maximum observed serum insulin icodec concentration after the last dose | From 0 to 168 hours after trial product administration (Day 36)
  hours
Terminal half-life for insulin icodec at steady state | Terminal part of the serum insulin icodec concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after last trial product administration (Day 36)
  hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (Dept.1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com